CLINICAL TRIAL: NCT03113526
Title: A Randomized Clinical Trial Comparing Output Volume Thresholds For Drain Removal After Selective Lateral Neck Dissections
Brief Title: Neck Drains for SLNDs
Acronym: SLNDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14209
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Neck Disease, Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Less than 30ml per 24-hour (Active Comparator): Drain removed as early as day one as long as output less than 30ml per 24-hour
  Interventions: Procedure: remove drain
- Less than 100ml per 24-hour (Active Comparator): Drain removed as early as day one as long as output less than 100ml per 24-hour
  Interventions: Procedure: remove drain

INTERVENTIONS:
Procedure: remove drain — remove drain when output is less than 30ml or less than 100ml per 24-hour

SUMMARY:
This is a single-blinded randomized controlled trial to compare the outcomes of early closed suction drain removal versus output volume-based drain removal after selective lateral neck dissections (SLND). The main hypothesis of the study is that the early drain removal of closed suction drains on the first postoperative day is safe compared to the current practice of output volume-based drain removal when output is less than 30ml/24hr or 15ml/12hr. This study will also evaluate the hypotheses that output volume-based drain removal of surgical drains increases inpatient length of stay and decreases the average patient satisfaction score on the measurement of quality of recovery (QoR-40).

DETAILED DESCRIPTION:
All adult patients (18 years old and over) undergoing unilateral SLNDs either levels I-III, I-IV, or II-III, II-IV, or II-VA for oral cavity, oropharynx (if the resection does not connect to the neck), thyroid, salivary gland, parotid, and skin carcinoma by one of three Head and Neck Surgery faculty members at UCSF will be consecutively registered. A randomized packet containing the patient's research ID number will be pulled and included into the patient's chart. Randomization will be done at the initiation of the study by creating a randomization list with blocking and stratification by surgeon. An envelope containing the patients randomized group assignment will not be opened until the end of the case. The patients will be randomized to one of two groups; drains placed routinely and removed once output is less than 30ml over 24-hours or 15ml over 12-hours and drains placed routinely and removed on rounds the morning of postoperative day one if output is less than 100ml total and does not appear chylous. Exclusion criteria will be bilateral neck dissections, revision neck dissections (prior surgery in the ipsilateral neck including excisional lymph node biopsy), previous radiation, need for sternocleidomastoid muscle (SCM) excision, need for internal jugular (IJ) excision, pectoralis major flap reconstruction of a ipsilateral skin defect, and anticoagulant medications other than routine deep venous thrombosis prophylaxis with either weight-based subcutaneous heparin or enoxaparin within 8 days postoperatively.

The procedure and postoperative care will be standardized to the degree described as follows: One 10 French Jackson-Pratt drain will be used. All necks will be closed with 3-0 vicryl, 4-0 monocryl, and 5-0 fast absorbing sutures. All patients will receive standardized postoperative orders including inpatient antibiotics not to exceed 24hrs (unless an infection is suspected) and deep vein thrombosis (DVT) prophylaxis; either weight based subcutaneous heparin or enoxaparin. The chief resident will receive an email indicating when to remove drain. All patients will receive standardized postoperative instructions including wound care with and without drain. A standardized physical exam will be performed on all patients every day of inpatient stay by the chief resident and on postoperative appointment (5-8 days post-operatively) by the attending surgeon to evaluate for clinical evidence of seroma and hematomas.

Physical exam will specifically include:

Inspect and palpate for presence fluctuance. Inspect for color change, erythema or ecchymosis Palpate for tenderness

All patients will be given a patient satisfaction questionnaire at their first postoperative visit to evaluate their overall satisfaction with their hospital stay, their recovery and healing of their wound, their comfort with home care, and level of pain. We plan to use the validated questionnaire, the measurement of quality of recovery (QoR-40).

Outcome Assessment: The primary outcome of this study will be the presence or absence of hematoma or seroma. Secondary outcomes will be the hospital length of stay, the need for any additional procedures, and the quantitative outcome from the patient satisfaction questionnaire. We will also collect data on the number of lymph nodes removed from the pathology report, the presence of carcinoma in the lymph nodes, and the need for home health care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing unilateral SLNDs either levels I-III, I-IV, II-III, or II-IV for oral cavity, oropharynx (if the resection does not connect to the neck), thyroid, salivary gland, parotid, and skin carcinoma.
2. A treatment plan involving levels I-III, I-IV, II-III, or II-IV, as recommended by National Comprehensive Cancer Network (NCCN) Guidelines
3. Patient must be 18 years of age or older.
4. The patient must have capacity to be able to sign a study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Pregnancy (for female patients).
2. Patients with history of prior radiation therapy or radioactive iodine to the head and neck.
3. Patients with neck dissection connected to upper aerodigestive tract.
4. Patients found to require sternocleidomastoid muscle or internal Jugular vein excision.
5. Patients who will require anticoagulant medications other than routine DVT prophylaxis within 8 days postoperatively
6. Patients undergoing bilateral neck dissection
7. Patients undergoing neck skin defect reconstruction
8. Patients with Chronic cough
9. Patients with bleeding disorders or who take aspirin regularly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Seroma formation | 30 days
  wound seroma

SECONDARY OUTCOMES:
Hospital length of stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: William Ryan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tamplen ML, Tamplen J, Shuman E, Heaton CM, George JR, Wang SJ, Ryan WR. Comparison of Output Volume Thresholds for Drain Removal After Selective Lateral Neck Dissection: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2017 Dec 1;143(12):1195-1199. doi: 10.1001/jamaoto.2017.1414. PMID 28837725